CLINICAL TRIAL: NCT03628066
Title: An Assessment of the Biological and Clinical Effects of Palbociclib (PD 0332991) With Ovarian Suppression and Letrozole in the Neoadjuvant Treatment of Patients With Premenopausal Estrogen-Receptor Positive/HER2-Negative Primary Breast Cancer
Brief Title: Biological and Clinical Effects of Palbociclib With Ovarian Suppression and Letrozole in the Neoadjuvant Treatment of Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Genomic Health®, Inc. (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-13
Record Dates: First submitted 2018-07-27; First posted 2018-08-14 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: Ovarian Suppression; Neoadjuvant; Premenopausal; Estrogen-Receptor Positive; HER2-Negative; Primary; Palbociclib; Letrozole; Goserelin; Ki67; Oncotype DX Breast Recurrence Score; Open-Label
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; palbociclib; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Oncotype DX Breast recurrence score on diagnostic tissue
  Daily Letrozole for 24 weeks + Palbociclib daily for 24 weeks + Goserelin weekly for 24 weeks
  Interventions: Drug: Letrozole; Drug: Palbociclib; Drug: Goserelin; Diagnostic Test: Oncotype DX Breast Recurrence Score

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5 mg by mouth daily for 24 weeks
  Other Names: Femara
Drug: Palbociclib — Palbociclib 125mg by mouth daily for 21 days per 28-day cycle (21 days on, 7 days off) for 24 weeks
  Other Names: Ibrance
Drug: Goserelin — Goserelin 3.6mg subcutaneous injection x 1 on Day 1 of each 28-day cycle for 24 weeks
  Other Names: Zoladex
Diagnostic Test: Oncotype DX Breast Recurrence Score — Prior to assignment to Arm 1 the Oncotype DX diagnostic test will be conducted on diagnostic tissue to assign a recurrence score for stratification to cohort 1 or 2.

SUMMARY:
This study will look at the safety and effectiveness of the combination of palbociclib and letrozole and ovarian suppression for premenopausal patients who have ER-positive/HER2-negative breast cancer that has not yet been treated.

DETAILED DESCRIPTION:
NSABP FB-13 is a phase II, open label study to examine the biological and clinical effect of neoadjuvant endocrine therapy with letrozole, palbociclib and ovarian suppression in premenopausal patients with estrogen-receptor (ER) positive, HER2-negative, early invasive breast cancer.

Premenopausal women newly diagnosed with ER-positive/HER2-negative early breast cancer who are suitable candidates for neoadjuvant endocrine therapy will be invited to join the FB-13 trial. A screening Oncotype DX Breast Recurrence Score® will be performed by Genomic Health, Inc. (GHI) on the diagnostic tissue of consenting patients to verify eligibility.

Patients will be stratified into one of two approximately equal sized cohorts based on baseline Breast Recurrence Score (RS) (cohort 1: patients with RS less than 11 or cohort 2: patients with RS 11 to less than 26).

Patients in both cohorts will receive letrozole 2.5 mg by mouth daily, palbociclib 125 mg by mouth daily for 21 days of a 28 day cycle, and goserelin 3.6 mg subcutaneous injection on Day 1 of each 28 day cycle. At Week 6 of study therapy, patients will have two core-cut biopsies. Patients from both cohorts who have a Ki67 less than 10% level will continue receiving study therapy for a total of 6 cycles. Patients with a persistent Ki67 greater than or equal to 10% at week 6 will permanently discontinue study therapy and begin neoadjuvant chemotherapy or proceed to surgery at the discretion of the treating physician.

Pre-treatment samples and post-surgical samples will be collected and analysed to identify subgroups of patients who may derive the most clinical benefit. The results of the biological analyses may allow a target sensitive population to be selected for future trials. The tissue collected in FB-13 will form an integral part of the primary analyses; so all core biopsies in this trial will be mandated for patients.

Two core-cut biopsies will be collected from each patient at baseline, after 6 weeks of study therapy, and upon completion of study therapy (24 weeks) at the time of definitive surgery.

Blood samples will be collected at baseline, 4 weeks, and at 24 weeks for estrone and estradiol levels to demonstrate ovarian suppression. A 4-week estradiol level in the postmenopausal range will be required to receive further treatment on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be premenopausal. Patients with a hysterectomy: menopausal status must be confirmed by estradiol and FSH.
* Operable hormonal receptor (HR) positive (ER/PR greater than or equal to 10%), HER2- negative, invasive early breast cancer, suitable for neoadjuvant AI treatment and ovarian suppression; HR- positive and HER2-negative as determined by American Society of Clinical Oncology/College of American Pathologists (ASCO-CAP ) guidelines.
* Diagnostic breast tissue must have an Oncotype DX Breast Recurrence Score® of less than 26 as determined by Genomic Health, Inc.
* No known severe hypersensitivity reactions to compounds similar to palbociclib or palbociclib excipients or to endocrine treatments.
* A breast tumor with an ultrasound size of at least 2.0 cm.
* Patients must have the ability to swallow oral medication.
* ECOG performance status of 0 or 1.
* At the time of randomization, blood counts performed within 2 weeks prior to randomization must meet the following criteria:

  * ANC must be greater than or equal to 1500/mm3
  * Platelet count must be greater than or equal to 100,000/mm3
  * Hemoglobin must be greater than or equal to 10g/dL.
* INR must be within normal limits of the local laboratory ranges. For laboratories that do not report an ULN for the INR assay, use less than or equal to 1.2 as the value for the ULN.
* The following criteria for evidence of adequate hepatic function performed within 2 weeks prior to study entry must be met:

  * Total bilirubin must be less than or equal to ULN for the lab unless the patient has a bilirubin elevation greater than ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and
  * Alkaline phosphatase must be must be less than or equal to 1.5 x ULN for the lab; and
  * AST and ALT must be less than or equal to 1.5 x ULN for the lab.
* Serum creatinine performed within 2 weeks prior to study entry must be less than or equal to 1.25 x ULN or estimated creatinine clearance greater than or equal to 60 mL/min (as calculated using the method standard for the institutions).

Exclusion Criteria:

* Active hepatitis B or hepatitis C with abnormal liver function tests.
* HIV positive patients receiving antivirals.
* Inflammatory/inoperable breast cancer.
* HER2-positive as determined using ASCO-CAP Guidelines.
* Oncotype Dx Breast Recurrence Score® result on diagnostic breast tissue greater than or equal to 26.
* Prior endocrine therapy for breast cancer.
* Any invasive malignancy within previous 5 years (other than basal cell carcinoma or cervical carcinoma in situ).
* Other nonmalignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow up such as:

  * Active infection or chronic infection requiring chronic suppressive antibiotics;
  * Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting gastrointestinal function;
  * Chronic daily treatment with corticosteroids with a dose of greater than or equal to 10 mg/day methylprednisolone equivalent (excluding inhaled steroids);
  * Seizure disorders requiring medication.
* Diagnosis by fine needle aspiration (FNA) alone or excisional biopsy or lumpectomy performed prior to study entry.
* Surgical axillary staging procedure prior to study procedure (with exception of FNA or core biopsy).
* Definitive clinical or radiologic evidence of metastatic disease.
* History of ipsilateral invasive breast cancer regardless of treatment or ipsilateral DCIS treated with radiotherapy or contralateral invasive breast cancer at any time.
* Any treatment, including radiotherapy, chemotherapy, and/or targeted therapy, administered for the currently diagnosed breast cancer prior to study entry.
* Use of any medication or substances that are strong inhibitors or inducers of CYP3A isoenzymes. Class III or Class IV myocardial disease as described by the New York Heart Association; a recent history (within 6 months) of myocardial infarction, or symptomatic arrhythmia at the time of randomization.

  * Class III: Patients with cardiac disease resulting in marked limitation of physical activity. Such patients are comfortable at rest. Less than ordinary physical activity that causes fatigue, palpitation, dyspnea, or anginal pain.
  * Class IV: Patients with cardiac disease resulting in inability to perform any physical activity without discomfort. Symptoms of cardiac insufficiency or anginal syndrome may be present even at rest.
* The investigator should assess the patient to determine if she has any psychiatric or addictive disorder or other condition that, in the opinion of the investigator, would preclude her from meeting the study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Complete Cell cycle arrest | From study entry to the time of the 6 week tumor biopsy to assess Ki67, approximately 6 weeks
  Percentage of patients with a Ki67 less than 2.7%

SECONDARY OUTCOMES:
Objective response rate | From study entry to the 24 week clinical assessment/ultrasound, approximately 24 weeks
  Objective response rate determined by breast tumor assessment measured by clinical exam and ultrasound
Pathologic complete response to study therapy (breast) | From study entry to time of surgery, generally 3 to 4 weeks after completion of study therapy at approximately 28 weeks
  Percentage of patients with absence of invasive cancer in surgical specimens
Pathologic complete response to study therapy (breast with nodes) | From study entry to time of surgery, generally 3 to 4 weeks after completion of study therapy at approximately 28 weeks
  Percentage of patients with absence of invasive cancer in surgical specimens
Correlation between Oncotype DX Breast Recurrence Score® and clinical Complete Response (cCR) | From study entry to the 24 week clinical assessment/ultrasound, approximately 24 weeks
  Correlation of the Oncotype DX Breast Recurrence Score® with clinical Complete Response
Correlation between Oncotype DX Breast Recurrence Score® and pathologic Complete Response (pCR) | From study entry to time of surgery, generally 3 to 4 weeks after completion of study therapy at approximately 28 weeks
  Correlation of the Oncotype DX Breast Recurrence Score® with pathologic Complete Response
Correlation between Oncotype DX Breast Recurrence Score® and Complete Cell cycle arrest rate (CCAR) | From the time of study entry to time of the 6-week tumor biopsy to assess Ki67, approximately 6 weeks
  Correlation of the Oncotype DX Breast Recurrence Score® with Complete Cell cycle arrest rate
Comparison between surgical intent and surgery received | From study entry to time of surgery, generally 3 to 4 weeks after completion of study therapy at approximately 28 weeks
  Changes between surgical intent declared at study start and actual surgery received after treatment
Comparison of estrone levels | From study entry to the 4 week blood draw, approximately 4 weeks
  Compare the estrone level at baseline to that after neoadjuvant treatment
Comparison of estradiol levels | From study entry to the 4 week blood draw, approximately 4 weeks
  Compare the estradiol level after neoadjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (15):
- United States (11):
  - Breast Cancer Care Specialist, Fountain Valley, California
  - Orange Coast Blood and Cancer Care, Fountain Valley, California
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Coast Hematology-Oncology Associates Medical Group, Long Beach, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Oncology Hematology Consultants, Long Beach, California
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Avera Cancer Institute-Sioux Falls, Sioux Falls, South Dakota
  - Lester and Sue Smith Breast Center, Houston, Texas
  - West Virginia University, Morgantown, West Virginia
  - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (4):
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - McGill University Health Centre-Cedars Cancer Centre, Montreal, Quebec
  - CHU de Quebec - Hopital de Saint-Sacrement, Québec, Quebec